CLINICAL TRIAL: NCT04890717
Title: Microbial Stool Biomarkers for Prediction of Autism and ADHD in Children
Brief Title: Biomarkers for Autism and ADHD in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: Mic_ASDADHD
Record Dates: First submitted 2021-05-09; First posted 2021-05-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Autism; ADHD
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ASD and/or ADHD children (Case group): Suspected or confirmed cases of ASD and/or ADHD children (Case group); no intervention(s) to be administered.
- Parent group: Parents of suspected or confirmed cases of ASD and/or ADHD children; no intervention(s) to be administered.
- Sibling group: Typically developed siblings of suspected or confirmed cases of ASD and/or ADHD children; no intervention(s) to be administered.
- Control group: Typically developed children not related to the case group ; no intervention(s) to be administered.

SUMMARY:
Autism (ASD) is one of the frequent neurodevelopmental disorders that children would occur. Many studies have shown that individuals with Autism are more common to experience significant gastrointestinal problems than other individuals. Symptoms include constipation, diarrhea, abdominal pain and gastric reflux. A recent study with 50 children with ASD, 50 children with other developmental disabilities and 50 healthy control children, it found that 70% of ASD children had presented with GI symptoms, compared with 42% of developmental disabilities children and 28% of developing children, it is believed that ASD children will have a distinctive microbial pattern in the stool.

Attention-deficit/hyperactivity disorder (ADHD) is another neurodevelopmental and neurobehavioral disorder. A study found that ADHD individuals experience significantly higher rate of stomach pain and bowel problems than other control individuals. It is suggested that the microbiota in the stool of ADHD children might be different. Genetic study also found that if a child has a sibling with ADHD, the risk of developing ADHD is three to four times higher than that of children with siblings without ADHD.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) was first developed by Kanner in 1943. In Hong Kong, a study showed that as many as 49 out of 10,000 children were diagnosed in Autism. ASD is one of the frequent neurodevelopmental disorders that children would occur. Many studies have shown that individuals with Autism are more common to experience significant gastrointestinal problems than other individuals. Symptoms include constipation, diarrhoea, abdominal pain and gastric reflux. In a study with 160 children with ASD, 59% had GI symptoms, including diarrhoea, unformed stool, constipation, bloating and gastroesophageal reflux (GERD). A study compared 51 ASD children, and 40 healthy control children found that 63% of ASD children had moderate or severe diarrhoea and constipation symptoms. In contrast, only 2% of control children had such experience. Similarly, a study of 150 children, with 50 children with ASD, 50 children with other developmental disabilities and 50 healthy control children, it found that 70% of ASD children had presented with GI symptoms, compared with 42% of developmental disabilities children and 28% of developing children. Other study stated that such untreated GI symptoms might worsen the behavioural issue of ASD children. As there is a strong relationship between ASD children and GI symptoms, it is believed that ASD children will have a distinctive microbial pattern in the stool.

Attention-deficit/hyperactivity disorder (ADHD) is another neurodevelopmental and neurobehavioral disorder. In Hong Kong, there were 8.9% of ADHD children among Primary one Chinese schoolboys. A large study (N=6483) found that ADHD individuals experience a significantly higher rate of stomach pain and bowel problems than other control individuals. McKeown did another study also reported that ADHD children were more likely to experience constipation and stool incontinence than normal healthy children. In one study that compared the Gastrointestinal Severity Index scoring between children with ADHD and healthy subjects, children with ADHD had significantly higher mean and scored higher in constipation, diarrhoea and flatulence variables. As the findings of ADHD individuals and gastrointestinal symptoms are closely associated, the microbiota in the stool might be different from normal children without ADHD.

Accumulating evidence implicated gut microbiota play a role in autism spectrum disorder (ASD). A huge community of microorganisms in the gastrointestinal (GI) tract impacts the development and function of the immune, metabolic, and nervous systems via the gut-brain axis. Majority of studies shown the diversity of gut microbiota changed in children with ASD compared with that of typically developing (TD) children, suggesting that the overall microbiota composition altered in ASD. Differences were observed between ASD and TD when comparing the abundance of bacteria in phyla and species level. Potential faecal bacteria biomarkers in the stool of children with ASD will be a useful non-invasive tool for early detection that will benefit more children with suspected conditions.

The microbiota was involved in many aspects of behaviour was confirmed in animal studies and human trial but it remains unclear whether gut microbiota recover in children with ASD after the intervention. Genetic research has revealed that if a child has a sibling with ADHD, the risk of developing ADHD is three to four times higher than that of children with siblings without ADHD.

Besides, previous studies showed that maternal unhealthy diet, tobacco use, and the harmful use of alcohol during pregnancy induce a shift in microbial ecology that negatively impacts offspring social behavior and has a fundamental role in the etiopathogenesis of ASD and ADHD. In some cases, children who have experienced stress, emotional abuse and violence are more prone to ADHD behaviour.

ELIGIBILITY:
Inclusion Criteria:

Case group, Sibling group and Control group:

* Children aged under 18 years old; and
* The parents or legal guardian agree to hand in the stool samples of children; and agree to complete questionnaires; and
* The parents or legal guardian agree to sign the informed consent form for the children

Parent group:

* Their suspected or confirmed ASD or ADHD children participated in the study; and
* Agree to hand in stool samples and complete questionnaires; and
* Agree to sign the informed consent consent

Exclusion Criteria:

All groups:

• Any subject taken probiotics, prebiotics, antibiotics 30 days before enrollment.

Subjects can be re-approached or join the study 30 days after taking probiotics, prebiotics, antibiotics.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects include
  * suspected or confirmed cases of ASD and/or ADHD children (Case group),
  * typically developed siblings of suspected or confirmed cases of ASD and/or ADHD children (Sibling group),
  * parents of suspected or confirmed cases of ASD and/or ADHD children (Parent group)
  * typically developed children not related to the case group (Control Group).
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-05-14 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify the microbial species in stool in suspected and confirmed ASD and/or ADHD children | 6 months
  Random Forest (RF) will be used for identifying the species of the biomarkers. The importance value of each species to the classification model will be evaluated by recursive feature elimination.

SECONDARY OUTCOMES:
To confirm different microbial species in stool in suspected and confirmed ASD and/or ADHD children across 2 years | 2 years
  Different species will be compared in terms of binary classifiers with Area Under the Curve (AUC) in Receiver Operating Characteristic (ROC) curves.
To confirm different microbial species in stool at different age groups in suspected and confirmed ADS and/or ADHD children across 2 years | 2 years
  Different species will be compared in terms of binary classifiers with Area Under the Curve (AUC) in Receiver Operating Characteristic (ROC) curves.
To correlate the changes in microbial species in stool with different diet habits in ASD and/or ADHD children across 2 years | 2 years
  Correlation statistical method will be used
To correlate the changes in microbial species in stool between the suspected and confirmed ASD and/or ADHD children with their siblings, parent or typically developed children at baseline | baseline
  Correlation statistical method will be used
To correlate the changes in microbial species in stool with different food additives levels in all subject groups at baseline | baseline
  Correlation statistical method will be used

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No